CLINICAL TRIAL: NCT05318937
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of SAGE-718 in Parkinson's Disease Cognitive Impairment
Brief Title: A Study to Evaluate the Effects of SAGE-718 in Participants With Parkinson's Disease Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 718-CNP-202
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Cognitive Dysfunction
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received SAGE-718-matching placebo, oral capsules, once daily (QD), in the morning for 42 days.
  Interventions: Drug: SAGE-718-matching placebo
- SAGE-718 (Experimental): Participants received SAGE-718, 1.2 milligrams (mg), oral capsules, QD in the morning for 42 days.
  Interventions: Drug: SAGE-718

INTERVENTIONS:
Drug: SAGE-718-matching placebo — Oral capsules
  Arms: Placebo
Drug: SAGE-718 — Oral capsules
  Arms: SAGE-718

SUMMARY:
The primary purpose of this study is to evaluate the effect of SAGE-718 on cognitive performance in participants with Parkinson's disease mild cognitive impairment (PD-MCI).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the following criteria for PD-MCI: Have a confirmed diagnosis of idiopathic Parkinson's disease (PD) according to 2015 Movement Disorder Society (MDS) clinical diagnostic criteria and meet MDS Task Force criteria for MCI in PD (excluding requirement for United Kingdom PD Brain Bank diagnostic criteria).
2. Meet the following criteria for Montreal Cognitive Assessment (MoCA): For participants meeting Level 1 PD-MCI criteria, have a MoCA score of 20 to 25 (inclusive) at Screening; For participants meeting Level 2 PD-MCI criteria (within the past year), have a MoCA score of 18 to 25 (inclusive) at Screening.
3. Meet criteria for modified Hoehn & Yahr Stage I to III (mild to moderate motor severity) at Screening.
4. Have stable motor symptoms for at least 4 weeks prior to Screening, in the opinion of the investigator.
5. Must be able to complete the Color Trails Test 1 (including the ability to follow rater redirection and correct errors), and, based on participant's performance and investigator's opinion, participant is expected to be capable of engaging in prolonged cognitive testing for the duration of the study.

Exclusion Criteria:

1. Have a diagnosis of dementia of any etiology, including but not limited to: Dementia with Lewy bodies, Alzheimer's dementia, and vascular dementia.
2. Have any parkinsonism other than PD, including secondary parkinsonism or atypical parkinsonism.
3. In the opinion of the investigator, be experiencing fluctuations in motor symptoms associated with PD that will interfere with completing study procedures.
4. Have an ongoing central nervous system condition other than PD that in the opinion of the investigator could influence the outcome of the study.
5. Have experienced significant psychotic symptoms, including hallucinations or delusions, within the past 3 months, in the opinion of the investigator.
6. Have a history of brain surgery, deep brain stimulation, or any history of hospitalization due to a brain injury.
7. Have a history, presence, and/or current evidence clinically relevant intracranial abnormality (e.g., stroke, hemorrhage, space-occupying lesion).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Sage Investigational Site, Sun City, Arizona
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, Fresno, California
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Los Angeles, California
  - Sage Investigational Site, Reseda, California
  - Sage Investigational Site, Sacramento, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Vernon, Connecticut
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Hialeah, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Port Orange, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Kansas City, Kansas
  - Sage Investigational Site, Bloomington, Minnesota
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Albany, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Stony Brook, New York
  - Sage Investigational Site, Williamsville, New York
  - Sage Investigational Site, Woodmere, New York
  - Sage Investigational Site, Raleigh, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Columbus, Ohio
  - Sage Investigational Site, Toledo, Ohio
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Nashville, Tennessee
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, San Antonio, Texas
  - Sage Investigational Site, Burlington, Vermont
  - Sage Investigational Site, Virginia Beach, Virginia
  - Sage Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 38 investigative sites in the United States from 06 June 2022 to 23 February 2024.
Pre-assignment Details: A total of 190 participants were screened, of which 86 participants were randomized to receive either SAGE-718 or placebo.
Period: Overall Study
Arm/Group | Placebo | SAGE-718
Started | 43 | 43
Completed | 42 | 39
Not Completed | 1 | 4
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants in the safety set (which included all participants who were administered at least one dose of the investigational product [IP]) who had baseline and at least 1 post-baseline efficacy evaluation.
Groups:
- Placebo: Participants received SAGE-718-matching placebo, oral capsules, QD in the morning for 42 days.
- SAGE-718: Participants received SAGE-718, 1.2 mg, oral capsules, QD in the morning for 42 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-718 | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (4.76) | 68.2 (6.37) | 68.3 (5.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 34 | 29 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 32 | 37 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 41 | 40 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding Test Score [Mean (Standard Deviation); unit: score on a scale] — The WAIS-IV coding test is a valid and sensitive measure of cognitive dysfunction that correlates with real-world functional outcomes (e.g., the ability to accomplish everyday tasks) and recovery from functional disability used to assess processing speed. The participant is required to identify the symbols matched to numbers using a key and write in the symbol beneath the associated number. The total score ranges from 0 to 135 and is based on the total number of codes correctly completed over a 120-second time limit. Higher scores indicate better processing speed. Population: Number analyzed is the number of participants with data available for analysis.
  score on a scale
    number analyzed (Participants) | 43 | 42 | 85
    (all) | 40.5 (13.27) | 39.7 (13.06) | 40.1 (13.10)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding Test Score
Description: The WAIS-IV coding test is a valid and sensitive measure of cognitive dysfunction that correlates with real-world functional outcomes (e.g., the ability to accomplish everyday tasks) and recovery from functional disability used to assess processing speed. The participant is required to identify the symbols matched to numbers using a key and write in the symbol beneath the associated number. The total score ranges from 0 to 135 and is based on the total number of codes correctly completed over a 120-second time limit. Higher scores indicate better processing speed. Positive change from baseline indicates better processing speed. Least Squares (LS) Means were calculated using a mixed-effects model for repeated measures (MMRM) approach.
Time Frame: Baseline, Day 42
Population: FAS included all participants in the safety set (which included all participants who were administered at least one dose of the IP) who had baseline and at least 1 post-baseline efficacy evaluation. Here, 'overall number of participants analyzed' signifies the number of participants with data available for analysis at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 42 | 40
score on a scale | 2.0 (1.44) | 2.0 (1.48)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.9934, MMRM — The p-value was obtained using a MMRM model which included treatment, visit, treatment-by-visit interaction as categorical covariates, and WAIS-IV at baseline as continuous covariates; Difference in LS Means = -0.0, 95% CI 2-sided [-4.13 to 4.09], Standard Error of Mean 2.07 — Difference was calculated as SAGE-718 - placebo

2. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as any AE on or after the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to Day 70
Population: The safety set included all participants who were administered at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 43 | 43
Participants | 27 | 21

3. Secondary Outcome: Number of Participants With at Least One TEAE by Severity
Description: A TEAE is defined as any AE on or after the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. Severity was assessed as:
  * Mild: symptoms barely noticeable to participant or does not make participant uncomfortable; does not influence performance or functioning; prescription drug not ordinarily needed for relief of symptoms
  * Moderate: symptoms of a sufficient severity to make participant uncomfortable; performance of daily activity is influenced; participant is able to continue in study; treatment for symptoms may be needed
  * Severe: symptoms cause severe discomfort; symptoms cause incapacitation or significant impact on participant's daily life; severity may cause cessation of treatment with IP; treatment for symptoms may be given and/or participant hospitalized.
  Participant with multiple instances of events is counted only once using maximum intensity.
Time Frame: Up to Day 70
Population: The safety set included all participants who were administered at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 43 | 43
Participants
  Mild | 15 | 14
  Moderate | 10 | 5
  Severe | 2 | 2

4. Secondary Outcome: Number of Participants Who Withdrew From Study Due to TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as any AE on or after the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to Day 70
Population: The safety set included all participants who were administered at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 70
Description: The safety set included all participants who were administered at least one dose of the IP.
Arm/Group | Placebo | SAGE-718
All-Cause Mortality (participants affected / at risk) | 1/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/43 | 3/43
Other Adverse Events (participants affected / at risk) | 4/43 | 5/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SAGE-718 (N=43)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SAGE-718 (N=43)
Urinary tract infection (Renal and urinary disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT05318937/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT05318937/SAP_001.pdf